CLINICAL TRIAL: NCT06987110
Title: A Randomized Clinical Trial Comparing Transverse Thoracic Plane Block, Midpoint Transverse Process Plane to Pleura Block and Erector Spinae Plane Block for Analgesia in Patients Undergoing Thoracoscopic Sympathectomy
Brief Title: Transverse Thoracic Plane Block, Midpoint Transverse Process Plane to Pleura Block and Erector Spinae Plane Block for Analgesia in Patients Undergoing Thoracoscopic Sympathectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdalsattar Elmohasseb, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1182/4/25.
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Transverse Thoracic Plane Block; Midpoint Transverse Process Plane to Pleura Block; Erector Spinae Plane Block; Analgesia; Thoracoscopic Sympathectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transverse thoracic plane block group (Experimental): Patients will receive a transverse thoracic plane block.
  Interventions: Other: Transverse thoracic plane block
- Midpoint transverse process plane to pleura block group (Experimental): Patients will receive a midpoint transverse process plane to pleura block.
  Interventions: Other: Midpoint transverse process plane to pleura block
- Erector spinae plane block group (Experimental): Patients will receive an erector spinae plane block.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Transverse thoracic plane block — Patients will receive a transverse thoracic plane block.
  Arms: Transverse thoracic plane block group
Other: Midpoint transverse process plane to pleura block — Patients will receive a midpoint transverse process plane to pleura block.
  Arms: Midpoint transverse process plane to pleura block group
Other: Erector spinae plane block — Patients will receive an erector spinae plane block.
  Arms: Erector spinae plane block group

SUMMARY:
This study compares the transversus thoracic muscle plane block (TTPB), midtransverse to pleura block (MTPB), and erector spinae plane block (ESPB) for postoperative analgesia in patients undergoing thoracoscopic sympathectomy.

DETAILED DESCRIPTION:
Thoracoscopic sympathectomy is a well-established procedure for the treatment of various hyperhidrosis disorders and certain vascular conditions, involving the division of sympathetic nerve fibers in the thoracic cavity.

The erector spinae plane block (ESPB) is an interfascial regional anesthesia block for thoracic analgesia which can be performed by superficial or deep needle approach.

The mid-transverse to pleura block (MTPB) was first described as a modified paravertebral block.

Transversus thoracic muscle plane block (TTPB) is a newly developed technique in which LA is injected into the fascial plane between the transversus thoracic muscle and the internal intercostal muscles for blocking the anterior cutaneous branches of intercostal nerves from thoracic (Th) 2 to Th 6.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for thoracoscopic sympathectomy

Exclusion Criteria:

* Coagulopathy.
* History of opiate abuse.
* Pre-existing chronic pain.
* Allergy to local anesthetics or analgesics.
* Infection at the site of injection.
* Mental or neurological disorders.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated)

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS)> 3 to be repeated after 30 min if pain persists until the VAS < 4
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of the surgery.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as pneumothorax, bradycardia, hypotension, nausea, vomiting, pruritis, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of the study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.